CLINICAL TRIAL: NCT04670237
Title: Clinical Outcome After Implantation of Medicontur Multifocal, Toric Intraocular Lens Liberty 677MTY: Rotational Stability, Visual Outcomes, Patients' Satisfaction, YAG Capsulotomy Rate
Brief Title: Clinical Outcome After Implantation of Medicontur Liberty 677MTY, a Multifocal, Toric IOL
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Medicontur Medical Engineering Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: MC_Liberty677MTY_HU_2019
Record Dates: First submitted 2020-12-10; First posted 2020-12-17 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Liberty677MTY Multifocal Toric IOL — multifocal, toric intraocular lens (IOL)

SUMMARY:
The purpose of this study is to evaluate visual outcomes, patient satisfaction and YAG capsulotomy rate after implantation of a multifocal toric lens- Liberty 677MTY - manufactured by Medicontur Ltd. (Zsámbék, Hungary),

DETAILED DESCRIPTION:
The purpose of this study is to evaluate visual outcomes, glass independency, visual disturbances (glares, halos), neuronal adaptation and patient satisfaction after implantation of multifocal diffractive apodized toric intraocular lens- Liberty 677MTY - diffractive-refractive apodized IOL based on EPS technology manufactured by Medicontur Ltd. (Zsámbék, Hungary).

The tested IOL model, Liberty 677MTY, has an overall length of 13 mm, an optic diameter of 6.0 mm without haptics angulations but with posterior vaulting. The refractive index of the optic material is 1.46 (at 23°C). The IOL is a single-piece-IOL, the optic and haptics are made from a hydrophilic acrylic co-polymer with integrated - covalently bound UV absorbent. The IOL is produced with yellow filter, covalently bound yellow chromophore. The toric component of Liberty 677MTY IOL is located on the posterior surface of the lens optic. The optic is marked with 2 marks. The marks are positioned exactly in middle between the two loops of haptic at the angulation at the flat axis of toric equivalent. The Liberty 677MTY is available with cylinder powers of 1.0 diopter (D) to 6.0 D. The IOL is designed with sharp edge following 360º to prevent migration of the lens epithelial cells , thereby to prevent PCO formation.

The trifocality of the lens is provided by the EPS technology recently developed by Medicontur uses an elevated phase shift on the central diffractive part of the lens in order to cause constructive interference between the 0th (far) and 1st diffractive (near) order, thus creating a 3rd (intermediate) focal point.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* astigmatism less than 1 dpt
* irregural astigmatism
* diabetic retinopathy
* iris neovascularisation
* serious intraoperative complications
* congenital eye abnormality
* glaucoma
* pseudoexfoliation syndrom
* amblyopia
* uveitis
* long-term anti-inflammatory treatment
* AMD (advanced AMD)
* retinal detachment
* prior ocular surgery in personal medical history
* corneal diseases
* severe retinal diseases (dystrophy, degeneration)
* severe myopia (if required IOL power is lower than 10 D)
* inadequate visualization of the fundus on preoperative examination
* patients deemed by the clinical investigator because of any systemic disease.
* eye trauma in medical history intraoperative exclusions:
* tear in capsulorhexis
* zonular dehiscence
* posterior capsular rupture
* vitreous loss and other unexpected surgical complication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The enrolled subjects will be the patients with cataract and pre-existing regular corneal astigmatism between 1.0 to 6.0 dpt. (Cylindric power of IOLs will range between 1.0 to 6.0 dpts). The patients will be indicated for cataract surgery and toric IOL implantation by the clinical investigator. The study will be conducted according to the tenets of the Declaration of Helsinki and patients will give informed consent after the nature and intent of study will be fully explained to them.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Rotational stability | 1 year
  Rotational stability will be measured using slit lamp images of the implanted lens on day one, seven, month one, three and one year postoperatively

SECONDARY OUTCOMES:
Visual outcome | 1 year
  Monocular and binocular visual aquity will be measured at far, intermediate and near by standard ETDRS chart at month one, three and one year postoperatively
Contrast sensitivity | 1 year
  Contrast sensitivity will be assessed by using the CSV-1000 method in photopic and mesopic light condition three month and one year after implantation
YAG capsulatomy | 1 year
  The rate of YAG capsulatomy will be assessed during the one year follow-up
Patient satisfaction | 1 year
  Patient satisfaction will be assessed by using the VFQ-25 questionnaire three month and one year postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Semmelweis University, Department of Ophthalmology, Budapest, Hungary